CLINICAL TRIAL: NCT00815412
Title: ACTIVATE: Standard Worksite Health Program vs. Activated Consumer
Acronym: ACTIVATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Paul E. Terry, PhD, President and Chief Operating Officer, StayWell
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01DP000104-03 (NIH)
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2008-12

CONDITIONS: Evidence of Improved Health Status
MeSH Terms: interventions — Counseling; Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Counseling in use of health care (Active Comparator)
  Interventions: Behavioral: Counseling in use of health care
- Counseling in diet, exercise (Active Comparator)
  Interventions: Behavioral: Counseling in diet, exercise
- Contol group (Placebo Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Counseling in use of health care
  Arms: Counseling in use of health care
Behavioral: Counseling in diet, exercise
  Arms: Counseling in diet, exercise
Other: Control
  Arms: Contol group

SUMMARY:
A 3-year, randomized, controlled trial comparing a traditional worksite health promotion program and an activated consumer program on health practices, health status and patient activation measures.

DETAILED DESCRIPTION:
The design is a cluster, randomized controlled trial of two companies with three arms in each company. The arms include two control groups (one from each company), two intervention groups using a standard health promotion intervention, and two intervention groups that constitute using an activated consumer intervention. The standard intervention includes educational offerings to address health behaviors. The activated consumer intervention offers shorter education sessions and includes decision tools and skills development for working with heath care providers to better manage health and clinical conditions. Variables include health risk assessments, clinical measures such as lipids, blood pressure, body mass index, and tobacco use, perception of health care consumer practices, claims costs, and absenteeism analysis.

ELIGIBILITY:
Inclusion Criteria:

* Airline and health care employees

Exclusion Criteria:

* Minors

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 2004-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Develop and evaluate a worksite-based, activated consumer intervention | March 2005; March 2007